CLINICAL TRIAL: NCT00243815
Title: Prophylactic Ibuprofen: Effect on IUD Continuation Rates
Brief Title: Use of Ibuprofen to Prevent IUD Site Effects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Chilean Institute of Reproductive Medicine (Other); Ministry of Health, Chile (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 9657
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2005-10

CONDITIONS: IUD Removal
Keywords: randomized controlled trial; prophylactic nonsteroidal antiflammatory drug; IUD removal
MeSH Terms: interventions — Ibuprofen

INTERVENTIONS:
Drug: ibuprofen

SUMMARY:
This research will determine whether prophylactic use of ibuprofen can prevent common side effects of the copper intrauterine device (IUD) and prevent early removal of the device.

DETAILED DESCRIPTION:
Increased menstrual bleeding and pain are the primary side effects that lead to early removal of the copper intrauterine device (IUD). Ibuprofen and other nonsteroidal anti-inflammatory drugs are a proven treatment for such IUD-induced problems. This study will determine if prophylactic use of ibuprofen can improve continuation rates of the IUD.

A total of 2,019 first-time IUD users were recruited in Chile for this double-blind, randomized, placebo-controlled trial. Half of the participants were given ibuprofen and instructions to take 1200 mg daily during menses (for up to 5 days each cycle) for the first six months of IUD use. The other half were asked to take an identical-appearing placebo in the same manner. The primary study endpoint was IUD removal within 12 months of insertion.

ELIGIBILITY:
Inclusion Criteria:

* mutually monogamous sexual relationship, less than 6 weeks since last menstrual period, more than six weeks since last pregnancy ended, residency within 50km of clinic, access to telephone, literacy

Exclusion Criteria:

* previous use of an IUD, history of liver and/or kidney disease, current of non-steroidal anti-inflammatory drugs, history of stomach ulcers and/or digestive hemorrhage, previous adverse reaction to ibuprofen and/or aspirin, symptoms of possible vaginal infection, current use of antibiotic or antifungal for genital tract infection, abnormal vaginal discharge, lesions in the vagina, known contraindication to IUD use, more than 3 alcoholic drinks per day

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2019
Dates: Start 2002-06; Study Completion 2004-11

PRIMARY OUTCOMES:
IUD removal

SECONDARY OUTCOMES:
Incidence of IUD side effects

CONTACTS AND LOCATIONS:
Overall Officials: David Hubacher, PhD, Principal Investigator — FHI 360
Locations (1):
- 43 Ministry of Health facilities, Santiago, Chile